CLINICAL TRIAL: NCT03861026
Title: Role of Cerebral Oximetry In Reducing Postoperative End Organ Dysfunction/Failure After Complex Non- Cardiac Surgery
Brief Title: Cerebral Oximetry to Reduce Organ Dysfunction After Non-cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-5747
Record Dates: First submitted 2018-05-15; First posted 2019-03-04 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Desaturation; Surgery

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomly allocated to either interventional or control groups according to a computer generated randomization code in predetermined size blocks.
  Bilateral NIRS (Masimo, O3TM Regional Oximetry) will be used to measure rSO2 intraoperatively.. The NIRS screen will be concealed in the control group to ensure blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Bilateral NIRS (Masimo, O3TM Regional Oximetry) will be used to measure rSO2 intraoperatively.
  In the interventional group, an alarm threshold at 90% of the baseline rSO2 value will be established. Based on predetermined algorithm the rSO2 will be maintained at or above 90% of the baseline measurements. The intervention will be commenced within 15 seconds of the reduction in rSO2 value.
  Interventions: Device: Bilateral NIRS (Masimo, O3TM Regional Oximetry)
- Control group (No Intervention): Bilateral NIRS (Masimo, O3TM Regional Oximetry) will be used to measure rSO2 intraoperatively.
  In the control group, the cerebral oximetry monitor screen will be concealed, however, the recording will be continuous after verification of the signal strength and baseline value by an independent observer trained in cerebral oximetry application and unaware of the study design.

INTERVENTIONS:
Device: Bilateral NIRS (Masimo, O3TM Regional Oximetry) — Bilateral NIRS (Masimo, O3TM Regional Oximetry) will be used to measure rSO2 intraoperatively. The NIRS electrodes will be placed on fronto-temporal area and baseline values of rSO2 obtained according to manufacturer's guidelines in the operating room prior to induction of anesthesia. The NIRS screen will be concealed in the control group to ensure blinding.
  Arms: Intervention group

SUMMARY:
Number of elderly patients requiring general anesthesia for major surgical procedures is increasing dramatically. It is estimated that 20% of these patients will develop major complications after surgery. Monitoring brain oxygen saturation may be helpful in reducing the postoperative complication rates. A decrease in brain oxygen is a sign that all other vital organs such as kidneys, heart, liver, and intestines have reduced blood supply and are starved from oxygen. This happens in 1 out of 5 patients undergoing major complex surgeries. Brain oxygen saturation monitor at this time is not used routinely during surgery, primarily due to the added cost, as well as, insufficient evidence that restoring the brain oxygen saturation to baseline would result in better outcomes. Patients will be randomly assigned to either study or control groups. In the study group, a special algorithm will be used to restore brain oxygen saturation. In the control group, the brain oxygen saturation will be monitored continuously, but the monitor screen will be electronically blinded, and standard clinical care applied. The objective of this study is to see if restoring the brain oxygen saturation to baseline results in less complication rates after surgery.

The objective of this study is to reduce the incidence of postoperative morbidity due to end organ dysfunction after major non-cardiac surgery in elderly patients.

The primary aim is to determine if restoration of rSO2 to baseline levels results in reduced incidence of major organ morbidity and mortality (MOMM).

A secondary aim is to determine a cost-effectiveness of this monitoring modality.

DETAILED DESCRIPTION:
The investigator will collect delirium, stroke, transient ischemic attacks, myocardial infarction (troponin essays), pulmonary embolism (clinical, echocardiography and computer tomography assessments), renal failure (creatinine increase by at least 50% from baseline), pneumonia (clinical, X-ray), atrial fibrillation (documented electrocardiogram), bleeding requiring a transfusion of more than or equal to 4 units of red blood cells within 72 hours of surgery, mechanical ventilation for 2 days, major wound disruption, surgical site infection, sepsis, septic shock, systemic inflammatory response syndrome (vasoactive medication requirement), unplanned return to the operating room, and vascular graft failure, for the duration of hospital stay, as well as, all-cause 30-day mortality. Frailty scale & DASI questionnaires will be administered at screening visit. Postoperative quality of recovery score (QoR-15) with be performed at baseline, POD 1 & 5 (discharge if earlier)]. Disability Free Survival (DFS) at 6 months (administer WHODAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients > 60 years of age
* Undergoing elective major non-cardiac surgery with an anticipated surgical duration of 4 hours or more,
* Preoperative written informed consent.

Exclusion Criteria:

* Emergency surgery
* Laparoscopic/Robotic surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
A composite outcome of major end organ dysfunction | surgery date to 6 months post surgery
  A composite outcome will be assessed as a dichotomous outcome. (YES or NO). All components of the composite outcome will be weighted equally. They will include the following outcomes: postoperative delirium assessed with Confusion Assessment Method (CAM), Stroke assessed clinically, Transient Ischemic Attacks assessed clinically, Myocardial infarction, Pulmonary Embolism, Renal failure, Pneumonia, Atrial fibrillation, bleeding, mechanical ventilation for ≥48 hours, Major wound disruption, Surgical site infection, Sepsis, Septic shock, Systemic inflammatory response syndrome, Vascular graft failure. Frailty scale & DASI questionnaires will be administered at screening visit.
  Postoperative quality of recovery score (QoR-15) with be performed at baseline, POD 1 & 5 (discharge if earlier)]. Disability Free Survival (DFS) at 6 months (WHODAS).

CONTACTS AND LOCATIONS:
Overall Officials: George Djaiani, Principal Investigator — Toronto General Hospital
Locations (2):
- Canada (2):
  - Tornoto General Hospital, University Health Network, Toronto, Ontario
  - Toronto General Hospital, Univerity health Network, Toronto, Ontario